CLINICAL TRIAL: NCT03521076
Title: Randomized Controlled Trial of Virtual Reality for Pain Management in a Specialty Rehabilitation Context
Brief Title: Randomized Controlled Trial of Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Chantel Burkitt, Clinical Scientist, Gillette Children's Specialty Healthcare
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: GilletteCSH
Record Dates: First submitted 2018-04-24; First posted 2018-05-11 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Muscle Spasticity
Keywords: Botulinum Toxin Injections; Virtual Reality
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Participants who are having botulinum toxin injections will be enrolled in the study. We will use a crossover study design, such that participants will access VR in addition to standard of care in one session and then experience only standard of care in the other condition. Participants will be randomized following the consent process. The participants will experience the opposite condition at their 2nd visit.
Who Masked: Outcomes Assessor
Masking Description: Researcher #1 will break the blind and know which condition the participant is in. Researcher #1 will then be the one to video record the treatment session. Researcher #1 will leave the room immediately following the treatment intervention. Researcher #2 will enter the room and will support the patient, parent/caregiver, and provider in completing outcomes assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual Reality for distraction (Experimental): The application of VR during the putative painful treatment (botulinum toxin injections) will provide a) active and engaging distraction during the procedure, and will b) block the view and auditory noise related to the procedure.
  Interventions: Device: Virtual Reality
- Standard of Care (No Intervention): Patients will receive the standard of care for the putative painful treatment (botulinum toxin injections).

INTERVENTIONS:
Device: Virtual Reality — Participants will have the opportunity to choose a game or relaxation experience to utilize during a botulinum toxin injection to distract from pain and anxiety during one visit. Virtual Reality will not be available during the other visit. AppliedVR has a number of games and relaxation experiences available for participants to chose from.
  Other Names: AppliedVR
  Arms: Virtual Reality for distraction

SUMMARY:
Measure pain and anxiety during a putative painful medical procedure (i.e., botulinum toxin injections) when Virtual Reality is employed compared to standard of care only using a Randomized Controlled Trial study design.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving botulinum toxin injections at Gillette Children's Specialty Healthcare

Exclusion Criteria:

* Patients who are fully anesthetized during their medical procedure
* Non-English speaking parents/patients
* Patients with history of motion sickness
* Patients with epilepsy
* Patients with a ventricular shunt
* Patients who have surgery during the study time period

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Faces Pain Scale - Revised (FPS-R) to assess intensity of pain during injections. | 2 days
  The Faces Pain Scale - Revised (FPS-R) will be used to assess pain intensity before, during, and after the treatment session. The FPS-R is a self-report measure of pain intensity developed for children. This scale shows a serious of six faces depicting increasing intensity of pain expression. The FPS-R instructions orient the child to the series of faces and then ask the child to point to the face that shows how much they hurt right now. Each face corresponds to a numerical rating between 0 and 10 (0, 2, 4, 6, 8, and 10). This rating scale corresponds to the widely accepted 0-to-10 metric for pain. The "0" equals no pain and the "10" equals very much pain. The score is reported as a total score.

SECONDARY OUTCOMES:
A series of visual analogue scales (VAS) to assess pain, anxiety, satisfaction with pain management, and perceived benefits of VR. | 2 days
  A visual analogue scale (VAS) will be used to quantify multiple aspects of the treatment experience expected to be impacted by the use of VR. The VAS will be a 10 cm 0-100 scale and will assess the following: patient anxiety before, during and after the procedure; parent/caregiver anxiety before, during, and after the procedure; proportion of the treatment time spent thinking about pain; worst pain during treatment; satisfaction with pain management; and nausea during treatment. This will be done at both visits (VR and no-VR).
Information collected from the medical record (e.g., medication use during procedure). | 2 days
  Following the signing of a HIPPA release, the medical record will be accessed to obtain such information as: patient diagnosis, date of birth, ethnicity, number of botulinum toxin injections, muscles injected, patient weight, height, and temperature, heart rate, blood pressure and oxygen saturation during treatment, clinical description of the context of VR use; provider description of whether VR enhanced clinical care; reduction or avoidance of medication due to VR; total amounts of medications given (e.g., valium, nitrous oxide, opioids; mg/kg); and notation of patient side effects from VR. This will be done at both visits (VR and no-VR).
The Pain Opinion Questionnaire (POQ) | 2 days
  The Pain Opinion Questionnaire (POQ) requires caregivers to respond to 5 questions in 3 separate sections regarding children with mild, moderate, and severe/profound intellectual and developmental disabilities. A description of the abilities and limitations of a typical individual with each level of impairment is provided in each section. The questions address 5 facets of pain: (a) the ability of the children to sense painful stimuli (Sensation), (b) how upset or distressed the children feel while in pain (Emotional Reaction), (c) how strongly the children react behaviorally to pain (Behavioral Reaction), (d) how much the children communicate their pain to others (Communication), and (e) how much pain the children suffer (Frequency). We are modifying the scale to require parents or caregivers to estimate whether they believe their child (not a hypothetical child) would experience that aspect of pain the "same as", "less than", or "more than" children without impairment.
The Dalhousie Pain Interview (DPI) | 2 days
  The Dalhousie Pain Interview (DPI) will provide a measure of pain experience in the previous week, including pain frequency (number of pain episodes), intensity (rated 0-10) and duration (number of seconds or minutes in pain). The measure consists of 10 items and was designed explicitly as an interview/survey script.
The Brief Pain Inventory (BPI) | 2 days
  The Brief Pain Inventory (BPI) will provide a measure of pain interference in the previous week (i.e., the degree to which ongoing pain interferes with daily living). The BPI is a 10-item, 11-point scale (0 = does not interfere, 10 = completely interferes). The items include general activity, mood, mobility, normal work, relationships with other people, sleep, enjoyment of life, self-care, recreational activities, and social activities. Total score (sum of all 12 items combined; range 0-120) and average score (average item score; range 0-10) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chantel Burkitt, PhD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- GilletteChildren's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breau LM, Burkitt C. Assessing pain in children with intellectual disabilities. Pain Res Manag. 2009 Mar-Apr;14(2):116-20. doi: 10.1155/2009/642352. PMID 19532853
- [Background] Vega-Avelaira D, McKelvey R, Hathway G, Fitzgerald M. The emergence of adolescent onset pain hypersensitivity following neonatal nerve injury. Mol Pain. 2012 Apr 24;8:30. doi: 10.1186/1744-8069-8-30. PMID 22531549
- [Background] Victoria NC, Inoue K, Young LJ, Murphy AZ. A single neonatal injury induces life-long deficits in response to stress. Dev Neurosci. 2013;35(4):326-37. doi: 10.1159/000351121. Epub 2013 Jul 5. PMID 23838073
- [Background] Santosh PJ, Baird G. Psychopharmacotherapy in children and adults with intellectual disability. Lancet. 1999 Jul 17;354(9174):233-42. doi: 10.1016/S0140-6736(98)07059-7. PMID 10421318
- [Background] Hoffman HG, Doctor JN, Patterson DR, Carrougher GJ, Furness TA 3rd. Virtual reality as an adjunctive pain control during burn wound care in adolescent patients. Pain. 2000 Mar;85(1-2):305-9. doi: 10.1016/s0304-3959(99)00275-4. PMID 10692634
- [Background] Sharar SR, Carrougher GJ, Nakamura D, Hoffman HG, Blough DK, Patterson DR. Factors influencing the efficacy of virtual reality distraction analgesia during postburn physical therapy: preliminary results from 3 ongoing studies. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S43-9. doi: 10.1016/j.apmr.2007.09.004. PMID 18036981
- [Background] Schmitt YS, Hoffman HG, Blough DK, Patterson DR, Jensen MP, Soltani M, Carrougher GJ, Nakamura D, Sharar SR. A randomized, controlled trial of immersive virtual reality analgesia, during physical therapy for pediatric burns. Burns. 2011 Feb;37(1):61-8. doi: 10.1016/j.burns.2010.07.007. Epub 2010 Aug 7. PMID 20692769
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Hua Y, Qiu R, Yao WY, Zhang Q, Chen XL. The Effect of Virtual Reality Distraction on Pain Relief During Dressing Changes in Children with Chronic Wounds on Lower Limbs. Pain Manag Nurs. 2015 Oct;16(5):685-91. doi: 10.1016/j.pmn.2015.03.001. Epub 2015 May 9. PMID 25972074
- [Background] Cacau Lde A, Oliveira GU, Maynard LG, Araujo Filho AA, Silva WM Jr, Cerqueria Neto ML, Antoniolli AR, Santana-Filho VJ. The use of the virtual reality as intervention tool in the postoperative of cardiac surgery. Rev Bras Cir Cardiovasc. 2013 Jun;28(2):281-9. doi: 10.5935/1678-9741.20130039. PMID 23939326
- [Background] Jones T, Moore T, Choo J. The Impact of Virtual Reality on Chronic Pain. PLoS One. 2016 Dec 20;11(12):e0167523. doi: 10.1371/journal.pone.0167523. eCollection 2016. PMID 27997539
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Steele E, Grimmer K, Thomas B, Mulley B, Fulton I, Hoffman H. Virtual reality as a pediatric pain modulation technique: a case study. Cyberpsychol Behav. 2003 Dec;6(6):633-8. doi: 10.1089/109493103322725405. PMID 14756928
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Ramstad K, Jahnsen R, Skjeldal OH, Diseth TH. Characteristics of recurrent musculoskeletal pain in children with cerebral palsy aged 8 to 18 years. Dev Med Child Neurol. 2011 Nov;53(11):1013-8. doi: 10.1111/j.1469-8749.2011.04070.x. PMID 22014321
- [Background] Hoffman HG, Patterson DR, Carrougher GJ. Use of virtual reality for adjunctive treatment of adult burn pain during physical therapy: a controlled study. Clin J Pain. 2000 Sep;16(3):244-50. doi: 10.1097/00002508-200009000-00010. PMID 11014398
- [Background] Sharar SR, Miller W, Teeley A, Soltani M, Hoffman HG, Jensen MP, Patterson DR. Applications of virtual reality for pain management in burn-injured patients. Expert Rev Neurother. 2008 Nov;8(11):1667-74. doi: 10.1586/14737175.8.11.1667. PMID 18986237
- [Background] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Background] Hoffman HG, Sharar SR, Coda B, Everett JJ, Ciol M, Richards T, Patterson DR. Manipulating presence influences the magnitude of virtual reality analgesia. Pain. 2004 Sep;111(1-2):162-8. doi: 10.1016/j.pain.2004.06.013. PMID 15327820
- [Background] Shinde SK, Danov S, Chen CC, Clary J, Harper V, Bodfish JW, Symons FJ. Convergent validity evidence for the Pain and Discomfort Scale (PADS) for pain assessment among adults with intellectual disability. Clin J Pain. 2014 Jun;30(6):536-43. doi: 10.1097/AJP.0000000000000020. PMID 24135902
- [Background] Breau LM, McGrath PJ, Camfield CS, Finley GA. Psychometric properties of the non-communicating children's pain checklist-revised. Pain. 2002 Sep;99(1-2):349-57. doi: 10.1016/s0304-3959(02)00179-3. PMID 12237214
- [Background] Phan A, Edwards CL, Robinson EL. The assessment of pain and discomfort in individuals with mental retardation. Res Dev Disabil. 2005 Sep-Oct;26(5):433-9. doi: 10.1016/j.ridd.2004.10.001. PMID 16039095
- [Background] Hoffman HG, Richards TL, Coda B, Bills AR, Blough D, Richards AL, Sharar SR. Modulation of thermal pain-related brain activity with virtual reality: evidence from fMRI. Neuroreport. 2004 Jun 7;15(8):1245-8. doi: 10.1097/01.wnr.0000127826.73576.91. PMID 15167542
- [Background] Wittwer A, Krummenacher P, La Marca R, Ehlert U, Folkers G. Salivary Alpha-Amylase Correlates with Subjective Heat Pain Perception. Pain Med. 2016 Jun;17(6):1131-6. doi: 10.1093/pm/pnv085. Epub 2016 Jan 13. PMID 26764337
- [Background] Norton M, Holm JE, McSherry WC 2nd. Behavioral assessment of relaxation: the validity of a Behavioral Rating Scale. J Behav Ther Exp Psychiatry. 1997 Jun;28(2):129-37. doi: 10.1016/s0005-7916(97)00004-9. PMID 9194010
- [Background] Barney CC, Krach LE, Rivard PF, Belew JL, Symons FJ. Motor function predicts parent-reported musculoskeletal pain in children with cerebral palsy. Pain Res Manag. 2013 Nov-Dec;18(6):323-7. doi: 10.1155/2013/813867. PMID 24308022
- [Background] Barney CC, Feyma T, Beisang A, Symons FJ. Pain experience and expression in Rett syndrome: Subjective and objective measurement approaches. J Dev Phys Disabil. 2015 Aug 1;27(4):417-429. doi: 10.1007/s10882-015-9427-3. Epub 2015 Mar 1. PMID 26425056
- [Background] Fernandez-Blazquez MA, Avila-Villanueva M, Lopez-Pina JA, Zea-Sevilla MA, Frades-Payo B. Psychometric properties of a new short version of the State-Trait Anxiety Inventory (STAI) for the assessment of anxiety in the elderly. Neurologia. 2015 Jul-Aug;30(6):352-8. doi: 10.1016/j.nrl.2013.12.015. Epub 2014 Jan 28. English, Spanish. PMID 24484757
- [Background] Perpina-Galvan J, Richart-Martinez M, Cabanero-Martinez MJ, Martinez-Dura I. Content validity of the short version of the subscale of the State-Trait Anxiety Inventory (STAI). Rev Lat Am Enfermagem. 2011 Jul-Aug;19(4):882-7. doi: 10.1590/s0104-11692011000400005. English, Portuguese, Spanish. PMID 21876939